CLINICAL TRIAL: NCT07255703
Title: Thoracic Surgery by SHURUI Single-Port Surgical Robot: A Prospective Single Centre Study
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Calvin Sze Hang Ng, Professor, Chinese University of Hong Kong
Other Study IDs: KF-600-3-583
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Thoracic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lobectomy, Segmentectomy Wedge resection of lung
  Interventions: Device: Device: Endoscopic Surgical System, SR-ENS-600
- Mediastinal Tumour Resection
  Interventions: Device: Device: Endoscopic Surgical System, SR-ENS-600

INTERVENTIONS:
Device: Device: Endoscopic Surgical System, SR-ENS-600 — undergoing robotic thoracic surgery by the Endoscopic Surgical System, SR-ENS-600

SUMMARY:
The introduction of single-port surgical robot has been a transformative breakthrough in the medical field, representing a significant advancement in minimally invasive procedures. One notable innovation is the SHURUI single-port surgical robot (SP), developed by Beijing Surgerii Robotics Company Limited. The SHURUI SP represents a cutting-edge technology in the field. This system features snake-like surgical instruments utilizing "dual continuum mechanism", which enables precise single-port procedures with wide range of motion and high load capacity.

The SHURUI SP has been cleared by the National Medical Products Administration (NMPA) of China for use in urology and gynecology and has completed clinical trials for general surgery and thoracic surgery. It is China's first and the world's second approved single-port surgical robot. Compared to multi-port surgical robots, it can provide patients with less trauma, fewer complications, and faster recovery.

The SHURUI SP has also achieved significant breakthroughs in clinical applications. It conducted the world's first randomized controlled clinical trial on single-port robotic urologic surgery and introduced a series of innovative surgical paradigms. These include the world's first single-port sleeve lobectomy, single-port retroperitoneal adrenalectomy, single-port retroperitoneal partial nephrectomy, single-port distal gastrectomy (Billroth I anastomosis), and single-port total gastrectomy.

Our centre is the first robotic surgical centre in Hong Kong since 2005. Over the years, we have established our centre to be one of the leading centre in Hong Kong and the region, with involvement in various new development in thoracic robotic procedures, publications and books, and more recently in robotic endo-lumenal procedures.

In this study, we evaluate the early surgical outcome and objective functional outcome of patients undergoing robotic thoracic surgery by SHURUI SP.

ELIGIBILITY:
Inclusion criteria:

1. Age between 18 - 75 years;
2. Subjects need to undergo endoscopic surgery and meet one of the following indications for surgical treatment:

   * Lobectomy, segmentectomy wedge resection of lung: Clinically diagnosed resectable early stage non-small cell lung carcinoma; oligometastatic cancer to the lung;
   * Mediastinal mass resection: Clinically diagnosed mediastinal tumour (benign or malignant) that are indicated for resection;
3. Preoperative ASA grade: Grade I-III;
4. Subject voluntarily participates in the clinical trial, and agrees or his/her guardian agrees and signs the informed consent.

Exclusion criteria:

1. Subjects with a previous history of thoracic surgery or other malignant tumor which, in the judgement of the investigator, make them unsuitable for enrolment;
2. Subjects with severe co-morbidities or organ dysfunction (heart, lung, liver, brain, kidney, etc.) or deemed too weak/ unsuitable for general anesthesia or operation;
3. Non-correctable coagulopathy and severe bleeding tendency；
4. Emergency surgery;
5. Severe obesity with BMI ≥30 kg/m2;
6. Subjects with severe allergic constitution, suspected or confirmed alcohol, drug addiction;
7. Other circumstances in which the investigator considered participation in this clinical trial inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Lobectomy, Segmentectomy, Wedge Resection of the lung, or Mediastinal Tumour Resection.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
conversion rate | 1 year + 1 month follow-up
  The feasibility of the Endoscopic Surgical System, SR-ENS-600 for thoracic robotic procedures (Lobectomy, Segmentectomy Wedge resection of lung and Mediastinal Tumour Resection), as measured by the conversion rate
major peri-operative complication rate (Clavein-Dindo grading III or above) | 1 year + 1 month follow-up
  The safety profile of the Endoscopic Surgical System, SR-ENS-600 for thoracic robotic procedures (Lobectomy, Segmentectomy Wedge resection of lung and Mediastinal Tumour Resection), as measured by the peri-operative complication profile.

SECONDARY OUTCOMES:
Operation time | 1 year
  The time from the beginning of the teleoperation to the ending of the teleoperation. Note: 1) the time of starting the skin incision, 2) the time of the surgical trolley parking, 3) the time of the positioning connection, 4) the time of starting teleoperation, 5) the time of finishing teleoperation, 6) the time of the closing skin incision.
  The operation-related time can reflect the maneuverability and ease of use of the instrument. Because the time of equipment preparation, skin incision, positioning connection and so on are interfered by many factors in the operating room, and the time from the beginning of teleoperation to the end of teleoperation is relatively stable, therefore, it is more objective to collect and analyze this period of time.
Estimated intraoperative blood loss (EBL) | 1 year
  Amount of intraoperative blood loss is recorded from the beginning to the end of the surgery
Length of hospital stay | 1 year + 1 month follow-up
  Total length of stay from the day of surgery to discharge. For subjects admitted in the afternoon/ discharged in the morning, 0.5 days were recorded on the day of admission/discharge.
Postoperative pain score | 1 year + 1 month follow-up
  time window: 24 ± 4 hours after surgery, 72 ± 4 hours after surgery, 120 ± 4 hours after surgery. This was assessed using the numerical rating scale (NRS) . The NRS score is clear and objective, which can help subjects make more accurate assessments and improve the comparability of assessments between different subjects. It was once considered the gold standard for pain assessment by the American Society of Pain[11]. This investigation used NRS versions 0-10, the most commonly used NRS (Figure. 5-1) . The subjects were assigned to 4 categories with 11 scores (0-10) : No Pain (0) , mild pain (1-3) , moderate pain (4-6) , and severe pain (7-10) . If the subject is discharged before a certain evaluation time point, the evaluation at that time point and after can not be carried out.
Blood transfusion rate | 1 year
  Proportion of subjects who underwent an intraoperative blood transfusion.
The Surgeon Satisfaction Questionnaire | 1 year+ 1 month follow-up
  time window: day 0 ~ within 24 hours after surgery. The Surgeon Satisfaction Questionnaire consists of two parts: the system (the"System" in this questionnaire refers to the investigational device "Endoscopic surgical system") performance-related (items 1 to 12, total of 12) and the surgeon comfort-related score (items 13 to 20, total of 8) . The Rating Scale: 5 points for each question, 1-5 points from top to bottom, full score of 100 points.
Perioperative complication | 1 year
  Surgical complication rates [ time window: within 30 ± 7 days after surgery] Possible intraoperative complications include thoracic adhesion, intraoperative bleeding, airway injury, and nerve injury. Possible postoperative complications include: pulmonary complications (including persistent air leak, pneumonia, atelectasis, pleural effusion, respiratory insufficiency/respiratory failure, etc.) , recurrent laryngeal nerve paralysis, chylothorax, etc.
device defects incidence | 1 year
  Incidence of device defects time window: the day of surgery. Device defect refers to the unreasonable risks that may endanger human health and safety, such as wrong label, quality problem, malfunction, etc.
readmission rate within 30 days after surgery | 1 month follow-up
  for operations other than segmentectomy/lobectomy reasons, not counted as reoperation rate
re-operation rate with 30 days after surgery | 1 month follow-up
  for reasons other than segmentectomy/lobectomy, not counted as the rate of reoperation
Mortality within 30 days after surgery | 1 month follow-up
  Mortality within 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Will need further discussion